CLINICAL TRIAL: NCT00560846
Title: Perioperative Nutrition in Upper GI Cancer Surgery (Oesophagectomy or Gastrectomy)
Brief Title: Perioperative Nutrition in Upper Gastrointestinal (GI) Cancer Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment over time.
Sponsor: Dan Azagury (Other)
Responsible Party: Sponsor-Investigator, Dan Azagury, Medecin adjoint du chef de service, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER: 07-123
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
Keywords: Gastric cancer; Esophageal cancer; Surgical complications; Immunonutrition
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition (Experimental): Pre-operative immunonutritrion, pre-operative glucose load, post-operative early immunonutrition
  Interventions: Dietary Supplement: Impact; Dietary Supplement: Glucose load
- Control (No Intervention): No immunonutrition, no glucose load, no early enteral immunonutrition

INTERVENTIONS:
Dietary Supplement: Impact — Preoperative 5 day oral Impact and early post-operative enteral Impact
  Arms: Nutrition
Dietary Supplement: Glucose load — Pre-operative glucose load: 800 ml of PreOp (Nutricia) 12 h before surgery; 400 ml of PreOp (Nutricia) 2 hours before surgery
  Other Names: PreOp Nutricia
  Arms: Nutrition

SUMMARY:
The aim of this study is to demonstrate the influence of peri-operative nutrition on the post-operative complications, preservation of lean body mass and length of stay after gastrectomy or oesophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for Upper GI cancer
* Age over 18
* Informed consent

Exclusion Criteria:

* Major swallowing disorders
* Dementia or other psychological state precluding compliance and understanding of research protocol
* Pre-existing enteral or parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative complications | 30 days
Length of stay | 30 days

SECONDARY OUTCOMES:
Quality of life | 1 year
Body composition | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dan E Azagury, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires Genève, Geneva, Canton of Geneva, Switzerland